CLINICAL TRIAL: NCT02643524
Title: Weight Change With Controlled Ankle Movement (CAM) Walker Boot Use
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: Nell Blake, DPM (Other)
Responsible Party: Sponsor-Investigator, Nell Blake, DPM, Assistant Professor, Department of Orthopaedics, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB - 2324
Record Dates: First submitted 2015-12-29; First posted 2015-12-31 (Estimated); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Foot Injury; Ankle Injury
Keywords: Adult; CAM boot; controlled ankle movement
MeSH Terms: conditions — Foot Injuries; Ankle Injuries | interventions — Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrition and Exercise Counseling (Active Comparator): CAM boot prescribed as standard of care Nutritional counseling provided Upper body exercise counseling provided Blood drawn for Albumin level at enrollment and final visit Height and weight measured at enrollment and final visit Patients in this arm compared with patients in control arm
  Interventions: Behavioral: Nutrition and Exercise Counseling
- Control (Active Comparator): CAM boot prescribed as standard of care No nutritional or exercise counseling provided Blood drawn for Albumin level at enrollment and final visit Height and weight measured at enrollment and final visit
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Nutrition and Exercise Counseling — Patients are prescribed CAM boot and provided nutritional and upper body exercise counseling at the time the CAM boot is dispensed. Patients will be given a diary to complete their daily meal intake (optional), seated upper body physical exercise guidelines and asked to perform them three days per week and each exercise three times per session if able. They will be asked to record number of hours CAM boot is worn daily in the Patient Diary, if one is utilized. Albumin lab test will be drawn and their height and weight measured.
  Arms: Nutrition and Exercise Counseling
Behavioral: Control — Patients are prescribed CAM boot. No nutritional or exercise guidelines will be provided. Patients will be given a diary to complete their daily meal intake and physician exercise (if any) and number of hours CAM boot is worn daily. Albumin lab test will be drawn and their height and weight measured.
  Arms: Control

SUMMARY:
The purpose of the study is to determine if patients wearing a CAM walker boot have a change in weight compared to patients who wear a CAM boot and are provided nutritional and upper body exercise information.

DETAILED DESCRIPTION:
The study objectives are: (1) Determine if patients wearing a CAM (Controlled Ankle Movement) walker boot have a change in weight compared to patients who wear a CAM boot and are provided nutritional and upper body exercises (gender appropriate) information at the time the CAM boot is dispensed; and (2) Determine, if weight is gained or lost, the average amount gained/lost over the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Age greater or equal to 18 (male or female)
* Participants prescribed a CAM boot as standard of care from the study investigator's practice
* Participant willing to have weight measured at the clinic site at time of enrollment and final visit
* Participants willing to have blood drawn for Albumin level at beginning and end of study
* Participant is able to provide voluntary, written informed consent
* Participant, in the opinion of the clinical investigator, is able to understand the clinical investigation and is willing to perform all study procedures and follow-up visits.
* Fluent in written and spoken English

Exclusion Criteria:

* Participants less than 18 years of age
* Pregnant women
* Cognitive impairment
* Participants with vertigo or other balance issues
* Participants unable to provide informed consent
* Non-English speaking individuals
* Participants who will not be wearing a CAM boot for at least 6 weeks
* Participants unable/unwilling to perform upper body exercises and follow nutrition guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-12-07 (Actual); Primary Completion 2018-04-09 (Actual); Study Completion 2019-05-23 (Actual)

PRIMARY OUTCOMES:
Weight change | Enrollment through release by Doctor to discontinue CAM Boot, an average of 12 weeks
  Determine weight gain or loss at time patient no longer is required to wear CAM boot, up to and including 12 weeks.

SECONDARY OUTCOMES:
Nutritional status (Pre- and post-albumin levels) | Enrollment through study completion, an average of 12 weeks.
  Pre- and post-albumin levels to measure protein and provide nutritional status

CONTACTS AND LOCATIONS:
Overall Officials: Nell Blake, DPM, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-30): https://cdn.clinicaltrials.gov/large-docs/24/NCT02643524/Prot_SAP_000.pdf